CLINICAL TRIAL: NCT04929535
Title: A Phase 2 Double-blind Placebo Randomized Controlled Trial of 30% Topical Application of Hydrogen Peroxide as Neoadjuvant Treatment of Non-melanoma Skin Cancers Prior to Definitive Surgery or Radiation
Brief Title: Hydrogen Peroxide Trial to Investigate the Efficacy of 30%H2O2 as a Topical Application Before Definitive Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JS10934
Record Dates: First submitted 2021-06-01; First posted 2021-06-18 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2021-08

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma of Skin Differentiated
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Hydrogen Peroxide; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30% hydrogen peroxide (Experimental): 30% hydrogen peroxide liquid topical application. 2 drops (0.10 ml) of hydrogen peroxide solution per centimeter of lesion. Once every week for continuous 4 weeks. If there is complete clinical response, further hydrogen peroxide will not be done.
  Interventions: Drug: Hydrogen Peroxide 30 % Topical Solution
- 3% hydrogen peroxide (Placebo Comparator): 3% hydrogen peroxide liquid topical application. 2 drops (0.10 ml) of hydrogen peroxide solution per centimeter of lesion. Once every week for continuous 4 weeks. If there is complete clinical response, further hydrogen peroxide will not be done.
  Interventions: Drug: Hydrogen Peroxide 30 % Topical Solution

INTERVENTIONS:
Drug: Hydrogen Peroxide 30 % Topical Solution — Patients will be seen by the radiation therapists involved with the study after randomization. Prior to application of hydrogen peroxide solutions, the patients' lesions will be prepared and debrided of keratinous debris and oils using sterile 70% isopropyl alcohol. Then, the appropriate hydrogen peroxide solution (30% for Arm 1 or 3% for Arm 2) will be rubbed into the lesion and a 1cm border all around the lesion until blanching of the lesion is observed. Hydrogen peroxide will be reapplied after one hour. This process will be repeated weekly for three additional applications for this study. If there is complete clinical response, further hydrogen peroxide will not be done. Patients will be accessed for definitive treatment 4 weeks later.
  Other Names: hydrogen peroxide

SUMMARY:
Previous work suggests that topical treatment with 33% hydrogen peroxide can reduce lesion size and, in about half of patients, can cause complete pathologic response. For patients with reduction in lesions size, the required size of the surgical excision or radiation field will be similarly decreased, thus potentially limiting associated morbidity and better cosmetic outcomes. Additionally, patients that experience a complete pathological response will be able to avoid additional treatment with either surgery or radiation. This will benefit both patients as well as helping to decreased use of health care resources. For the current study we will be using 30% hydrogen peroxide as it is commercially available. If this study shows positive results, it could lead to significant benefit on both a patient and systems level. Locally, our cancer Centre treats approximately 700 new patients per year who fit into the study criteria and could potentially benefit from this novel neoadjuvant treatment that is fairly inexpensive.

DETAILED DESCRIPTION:
Non-melanoma skin cancers (NMSC) are the most commonly occurring cancers worldwide and the incidence of these malignancies is steadily rising secondary to the advancing age of the general population as well as sun exposure. Gold standard treatment modalities for NMSC include surgical excision and radiation therapy. Both of these treatments are accompanied by risks to the patient including pain, bleeding, infection, scarring and pigment alterations. Larger lesions necessitate treatment of larger areas of skin, which can worsen treatment related toxicities. Patients with NMSC of the head and neck may be particularly concerned regarding these risks as this region is cosmetically sensitive.

For surgery, a recommended margin of 0.5-1.0cm of normal tissue is removed beyond the lesion boarder to decrease risk of recurrence. In an area like the face, reconstruction of excision defects and ultimately aesthetic outcomes are of utmost importance. Particularly large skin can sometimes necessitate rotational flaps or even skin grafting, both of which have drawbacks in terms of healing, scarring, and surgical complications. A similar issue of margins arises with radiation. For patients undergoing radiation treatment with an orthovoltage a margin of 1.0cm is added beyond the clinical boarders of the lesion, while for patients being treated on an electron unit, a 1.5cm margin is added.

Currently, there are no routinely used neoadjuvant treatment option that can be used to help decrease lesion size and therefore limit toxicities associated with definitive treatment (surgery or radiation). However, these has be recent work looking at neoadjuvant use of concentrated hydrogen peroxide in reduction of lesion size (5).

Hydrogen peroxide a product of respiration in mitochondria and an important oxidizing agent in biological system. As it is a potent oxidizing agent, hydrogen peroxide can exert a role in oxidative stress, although the exact mechanism through which this occurs is not yet known. Giulivi and Davies (1) propose that hydrogen peroxide may interact with hemoglobin in the dermal capillaries producing oxidized forms of hemoglobin such as ferryl hemoglobin which is highly reactive. It is therefore possible that hydrogen peroxide could cause necrogenous oxidation and oxygen induced apoptosis of cells in NMSC.

Dilute hydrogen peroxide it is used frequently as a topical antiseptic and hemostatic agent (2). These effects are generally achieved with topical application of 3% hydrogen peroxide to the skin, with little to no side effects for patients aside from some mild discomfort. As far as potential clinical application of more concentrated hydrogen peroxide, a previous investigation examining the use of hydrogen peroxide at or above a concentration of 23% in the treatment of seborrheic keratosis found that the mean number of benign lesions remaining 90 days after treatment was significantly lower in the hydrogen peroxide group compared to placebo (3). The average number of applications of hydrogen peroxide was 6, separated by approximately one-week intervals (3). In this study, the only side effect from application of the hydrogen peroxide solution was less than ten minutes of "burning" at the application site (3). Hydrogen peroxide has also been used in combination with other topical treatments such as non-steroidal anti-inflammatories (NSAIDs) to successfully combat precancerous lesions such as actinic keratosis (4) as well as part of photodynamic therapy protocols in the treatment of skin cancers.

Recently Mundi et al. (5) published a case series looking at the role of a topical application of 33% hydrogen peroxide as neoadjuvant therapy before surgical excision. This series included 11 patients and a total of 17 lesions. Patients received multiple topical applications of hydrogen peroxide and were evaluated 4 weeks after the initial treatment to assess response. There was complete pathological response in 53% of patients and the remained had a statistically significant reduction in the size of the lesion requiring a smaller surgical excision. Although promising, this was a small, non-randomized, non-controlled proof of concept study. Further work is required before this type of treatment could be adopted commonly or used of trial.

However, given its relatively benign nature and previous efficacy in treating other skin growths, hydrogen peroxide may represent a simple yet effective method at shrinking NMSC of the head and neck before they are excised or radiated. In doing so, it could minimize the invasiveness of surgical excision thereby accelerating healing and improving aesthetic outcomes for patients. If patients are being treated with radiation, we may be able to use smaller radiation fields with less side effects, better cosmesis and improved local control.

This double-blind placebo randomized controlled trial will seek to investigate the role of neoadjuvant hydrogen peroxide prior to definitive treatment with either surgery or radiation. For the purposes of this trial a concentration of 30% hydrogen peroxide will be used as this is the highest concentration easily available.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed measurable basal cell carcinoma (BCC) or well to moderately differentiated squamous cell carcinoma (SCC)
* Age 18 years or older
* Able to provide informed consent

Exclusion Criteria:

* Lesion with indistinct borders
* Any evidence of metastatic disease
* Poor performance status (Eastern Cooperative Oncology Group > 1) with life expectancy of less than 2 years
* Gorlins syndrome, a genetic predisposition to multiple skin cancers where surveillance and early intervention is of paramount importance
* Any recurrent cancer after surgery or radiation
* Very extensive carcinoma that cannot be readily removed by surgery or treated by radiation using orthovoltage or electron beam
* History of cutaneous photosensitization, porphyria or photodimerization as their tolerance to hydrogen peroxide application is unpredictable
* Previous application of 5-Fluorouracil cream to the lesion within the last 8 weeks
* Any immune-compromised patients where skin cancers can be very aggressive
* Patients who are unwilling to return for 1-year follow-up assessment
* Poorly differentiated SCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in lesion size | 4 weeks after the last application of hydrogen peroxide
  Reduction in lesion size, measured in square centimeter, 4 weeks after the last application of hydrogen peroxide.

SECONDARY OUTCOMES:
Proportion of Patients with complete response | At study completion, an approximate of 1 year
  Proportion of patients with complete response not requiring surgery or radiation.
Proportion of patients requiring definitive surgery | At study completion, an approximate of 1 year
  Proportion of patients requiring definitive surgery or radiation who achieve complete clinical response, but not complete pathological response following hydrogen peroxide treatment.
Size of surgically removed skin | At study completion, an approximate of 1 year
  Reduction in the size of the skin, measured in square centimeter, that needs to be surgically removed before and after hydrogen peroxide treatment for patients selecting surgery
Change in the size of the radiation field | At study completion, an approximate of 1 year
  Reduction in the size of the radiation field, measured in square centimeter, before and after hydrogen peroxide treatment for patients selecting radiation.
Local Control | At study completion, an approximate of 1 year
  Clinical local control at one year after randomization.
Adverse Events | At baseline, week 1, week 2, week 3, and also at 4 weeks after last hydrogen peroxide application. Adverse events will also be assessed at 3, 6, 9 and 12 months after the baseline visit.
  Adverse events associated with hydrogen peroxide treatment, assessed using standardized questionnaire one week after each application. Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life-threatening or disabling, Grade 5: Death.

CONTACTS AND LOCATIONS:
Overall Officials: Jinka Sathya, MD, Principal Investigator — Western University
Locations (1):
- London Regional Cancer Program, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No